CLINICAL TRIAL: NCT07184762
Title: Clinical, Radiographic and Histological Evaluation of Z-shaped Bone Plates in Management of Mandibular Fractures
Brief Title: Evaluation of Z-shaped Bone Plates in Management of Mandibular Fractures
Acronym: z-FIX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Eman Mohamed Eldemardash Ali, Assistant Lecturer oral and maxillofacial surgery department, Faculty of Dentistry, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 657\2023
Record Dates: First submitted 2025-09-04; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mandibular Fracture Treatment
Keywords: mandibular fracture; open reduction; z-shaped plate; conventional bone plates
MeSH Terms: conditions — Mandibular Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal; Bone Plates

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- z-plate (Experimental): mandibular fracture will be reduced and fixed with Z shaped bone plate
  Interventions: Procedure: open reduction and internal fixation with bone plate; Procedure: z-plates.
- conventional Miniplate (Active Comparator): mandibular fracture will be reduced and fixed with conventional two miniplates.
  Interventions: Procedure: open reduction and internal fixation with bone plate; Procedure: conventional miniplates.

INTERVENTIONS:
Procedure: open reduction and internal fixation with bone plate — mandibular fracture were reduced and fixed with bone plates.
Procedure: z-plates. — mandibular fracture were reduced and fixed with z-plate miniplates.
  Arms: z-plate
Procedure: conventional miniplates. — mandibular fracture were reduced and fixed with conventional two miniplates.
  Arms: conventional Miniplate

SUMMARY:
he goal of this clinical trial is to evaluate Z shaped bone plate in mandibular fracture treatment regarding post operative healing, function restoration and esthetic.

aims to answer are: In mandibular trauma population, what is the difference between internal fixation using conventional miniplates compared to z shaped bone plates regarding post operative healing, function restoration and esthetic?

Participants will be divided equally and randomly in 2 groups as follows:

Group A: eight patients treated with Z shaped bone plate. (Study group) Group B: eight patients restored with conventional two miniplates.(control group)

DETAILED DESCRIPTION:
Introduction: Various miniplate systems have been developed in recent years including three-dimensional miniplate, microplates and bioresorbable plate, and their advantages and disadvantages have been compared and studied. To overcome the shortcomings of 3D plating system such as difficulty in adaptation and fixation in fractures involving the mental nerve, a Z plate has been designed. Aim: to evaluate Z shaped bone plates in mandibular fracture management clinically, radiographically, and histologically. Methodology: sixteen patients with mandibular fracture grouped to two groups group A managed by Z plates, group B managed by two miniplates. Patients will follow up clinically postoperative. Radiographic evaluation will be performed immediately postoperative, 1 month and 4 months Experimental study will be on dogs and histological evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are suffering from recent, uninfected, and minimally displaced or unfavorable fractures at the symphysial or parasymphysis region of the mandible.
2. Adult patients with no gender predilection that agreed to present for follow-up visits for minimum postoperative period of immediate, month, 3 months,6 months.
3. A fracture that demands open reduction and internal fixation
4. Medically fit patients for general anesthesia

Exclusion Criteria:

1. Comminuted, infected mandibular fracture.
2. Pediatric patients below 14 years of age
3. geriatric patients with completely edentulous mouth.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Radiographic evaluation (Bone density ratio at fracture line ) measured using orthopantomograms (OPGs) by ImageJ software. | within 1week postoperative, 1month, 4month
  Radiographic evaluation using orthopantomograms (OPGs) is performed immediately postoperatively, at 1 month and 4 months.
  To assess bone density along the fracture line, a densitometric analysis was conducted using the ImageJ system.
  Digital images are analyzed using ImageJ software. The mean gray value of a region of interest (ROI) drawn along the entire length of the fracture line was calculated. This gray value represents the relative bone density within the fracture site. Range: 0.0 - 1.0 (unitless ratio).
  Higher values indicate greater bone density and better healing
Postoperative pain assessed using the Visual Analog Scale (VAS) | day 1 , day 3, and 1week postoperative
  postoperative pain assessed using the Visual Analog Scale (VAS). Range: 0 (no pain) - 10 (worst imaginable pain). Higher scores indicate worse pain

SECONDARY OUTCOMES:
Clinical fracture stability evaluated by manual mobility test and tenderness on palpation. | 1 week postoperative,1month, 3 months, 6 months
  Outcome: Stable vs. unstable fracture (binary measure) assessed through bimanual digital manipulation i. Stable >> no movement of fragments. ii. Nonstable>> presence of movement

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S. Hamed, professor, Study Chair — Oral and Maxillofacial Surgery, Faculty of Dentistry, Suez Canal University; Mohamed A. Elsholkamy, professor, Study Director — Oral and Maxillofacial Surgery, Faculty of Dentistry, Suez Canal University; Amr A. Gomaa, associate professor, Study Director — plastic Surgery, Faculty of medicine, Suez Canal University; Eman M. Eldemardash, assistant lecturer, Principal Investigator — Oral and Maxillofacial Surgery, Faculty of Dentistry, Suez Canal University
Locations (1):
- Suez Canal University hospital, Ismailia, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No